CLINICAL TRIAL: NCT05526963
Title: Reduction of Polypharmacy in Elderly People With Multiple Diseases - a Stepped Wedge Cluster-randomized Controlled Trial
Brief Title: Reduction of Polypharmacy in Elderly People With Multiple Diseases
Acronym: RED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: University of Leipzig (Other); Hannover Medical School (Other)
Responsible Party: Principal Investigator, Alexander Bauer, Reserach Coordinator, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RaPHaeL_001_RED
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Polypharmacy; Multimorbidity
Keywords: Primary Care; Polypharmacy; Multimorbidity; Drug-Related Side Effects and Adverse Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster-randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Medication review (STOPP/START-criteria) + telephone-based adherence support measure (motivational interviewing)
  Interventions: Other: Medication plan review; Behavioral: Adherence support
- Control Group (No Intervention): Usual care

INTERVENTIONS:
Other: Medication plan review — Intervention group patients will receive a revised medication plan by external pharmacologist based on the the STOPP/START criteria. The revised medication plan will be provided to the family physician who then will provide it to the patient. The revision comes along with evidence based information for the physician to prevent possible uncertainties by the physicians.
  Arms: Intervention Group
Behavioral: Adherence support — Intervention group patients will receive a study nurse administered adherence support measure based on telephone-based motivational interviewing. The measure includes information on possible consequences of inadherence and signs of adverse drug reactions that is comprehensible for lay persons.
  Arms: Intervention Group

SUMMARY:
Elderly GP patients are often treated with five or more medications and therefore prone to adverse drug reactions (ADR). Potentially inappropriate prescriptions (PIPs) lead to increased adverse events like falls, hospitalizations and mortality. The primary aim of this study to reduce the frequency of ADRs in multimorbid patients aged 70 years and older by reducing polypharmacy.

DETAILED DESCRIPTION:
Introduction: Many elderly people are multimorbid and are treated with five or more medications (polypharmacy) at the same time. Due to age related physiological changes they are especially vulnerable to adverse drug reactions (ADR). Potentially inappropriate prescriptions (PIPs) lead to increased adverse events like falls, hospitalizations and mortality. Up to 16% of unplanned hospitalizations of elderly people with polypharmacy are caused by ADRs. The primary aim of this study is the evaluation of the effectivity of a multi-component-intervention to reduce the frequency of ADRs in multimorbid patients aged 70 years and older.

Methods: We are planning a multi-center stepped wedge cluster randomized controlled trial at 40 primary care practices affiliated to the RaPHaeL-network (Research Practices Halle-Leipzig) in Saxony-Anhalt and Saxony, Germany. The planned intervention follows the recommendations of the New Medical Research Council and comprises a pharmacological medication plan review according to the STOPP/START-criteria and an adherence support measure employing motivational interviewing. Control group will receive usual care. Eligible patients are ≥ 70 years old, are diagnosed with three or more chronic medical conditions and are prescribed five or more medications. The primary outcome is the rate of ADRs six months post intervention. The secondary outcomes are number of ADRs, hospitalization rate due to ADRs, medication adherence (Morisky Adherence Score MMAS-8), the health-related quality of life (Euro-QOL EQ-5D-5L), the number of PIPs (according to STOPP/START), number of primary care physician per quarter, the medication appropriateness index and the mean number of de-prescriptions per patient. The planned sample size is 1,146 patients.

Discussion: Multimorbid patients with polypharmacy show an increased risk for PIPs, since prescriptions can be based on evidence for pharmacological therapy of a single condition without taking into account the complex drug interactions. Based on the existing evidence we are aiming to reduce ADRs in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 5 longterm medications (> 6 months) (polypharmacy)
* ≥ 3 chronic diseases (multimorbidity)
* ≥ 1 family doctor consultation within the last 6 months

Exclusion Criteria:

* Patients with a critically reduced life expectancy
* Patients who cannot autonomously visit the family practice
* Patients who cannot participate in the informed consent process
* Patients who are residing in a nursing home
* Patients with dementia or a mental of behavioral disorder ICD-10 F00-F99
* Patients who are participating in another medical study with a focus on polypharmacy or multimorbidity

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1146 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse drug reactions | 6 months
  Rate of self-reported adverse drug reactions per patient based on a list of commonly reported drug-related symptoms in primary care.

SECONDARY OUTCOMES:
Potentially inappropriate prescriptions | 6 months
  The number of potentially inappropriate prescriptions based on the STOPP(Screening Tool of Older Persons' potentially inappropriate Prescriptions) and START (Screening Tool to Alert doctors to Right Treatment) criteria.
Hospitalizations | 6 months
  The frequency of hospitalizations due to adverse drug reactions.
Adherence | 6 months
  The patient's adherence to the medication plan based on the Morisky medication adherence score 8 (MMAS-8). Response categories are yes/no for each item with a dichotomous response and a 5-point Likert response for the last item. The summed total score ranges from 0 to 8 otal MMAS-8 scores can range from 0 to 8 and will be been categorized into three levels of adherence: high adherence (score = 8), medium adherence (score of 6 to < 8), and low adherence (score< 6).
Health-related quality of life | 6 months
  The health-related quality of life will be measured using the six-item European Quality of Life 5 Dimensions 3 Level Version (Euro-QOL EQ-5D-5L) tool, ranging from 0 to 100 on a visual analoge scale with higher values indicating a higher quality of life.
Family doctor consultations | 6 months
  The number of family doctor consultations within the time frame between recruitment and follow-up.
Medication appropriateness | 6 months
  The medication appropriateness will be measured using the medication appropriateness index (MAI)
Deprescription | 6 months
  The number of medication de-prescriptions per patient
Types of adverse drug reactions | 6 months
  Number and types of self-reported adverse drug reactions per patient based on a list of commonly reported drug-related symptoms in primary care. Each symptom's severity will be quantified by use of an analogue scale from 0 (no severity) to 10 (maximum imaginable severity)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frese, Prof., Study Chair — MLU Halle-Wittenberg
Locations (1):
- HAP ANZ, Halle, Saxony-Anhalt, Germany